CLINICAL TRIAL: NCT03951428
Title: Screening and Early Detection of Cancer Through Identification of Novel Female Specific Biomarkers Through Self-Collected Menstrual Blood
Brief Title: Screening of Cancer Through Novel Female Specific Biomarkers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: LifeStory Health Inc. (Industry)
Collaborators: Baylor Scott and White Health (Other)
Responsible Party: Sponsor
Other Study IDs: LSHBSWMBC
Record Dates: First submitted 2019-05-13; First posted 2019-05-15 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- All Participants
  Interventions: Diagnostic Test: Menstrual Blood Screening Test

INTERVENTIONS:
Diagnostic Test: Menstrual Blood Screening Test — The sponsor will be testing women's menstrual blood to investigate the feasibility and efficacy of assessing three early stage cancers via self-collected menstrual blood using FDA approved devices.

SUMMARY:
Can reliable biomarkers be identified for detection of cancer at early stages using menstrual blood (MB)? Preliminary mass spectrometry (MS) results suggest that MB provides biomarkers for identification of disease such as cancers.

DETAILED DESCRIPTION:
The sponsor will first analyze menstrual blood (MB) samples in three discreet studies: breast, endometrial, lung. According to American Institute for Cancer Research, "Endometrial cancer is the most common cancer of the female reproductive organs. More cases of endometrial cancer occur each year than ovarian and cervical cancers combined." 20% to 25% will be diagnosed with endometrial cancer before menopause. Based on the patient recruitment potential and high impact on women's health, these three cancer types are suitable models to evaluate the expediency of utilizing MB as an ideal source for identification of cancer markers.

Health profiles are completed by all participants and where applicable and possible, patient medical records, health tracking device data, etc. will be included. Blood samples will be collected as indicated on the collection protocol outlined by LifeStory Health's (LSH's) Protocol and Instructions for Use. Samples will be collected in the participant's home according to LSH's Collection Protocol using EBF-Inc.'s 903 dried blood spot (DBS) collection device prior shipment to the research center. Samples should be sent within 3 days of collection. Up to one-hundred and fifty micro-liters (150 uL) of menstrual blood can be collected from donors using the collection device.Samples will be processed according to LSH's protocol and any methods outlined in this development plan.

The study will receive samples from 60 female participants, totaling 30 samples from early-stage cancer patients and 30 samples from healthy women. After initial determination of potential cancer markers for all three cancer types, the sponsor will select a single cancer type with the most promising results ("Cancer 1") and carry out additional, statistically higher-powered, studies on all four stages of this selected cancer. After the identities of potential MB biomarkers for a single cancer type are re-confirmed and established at the highest level of confidence, simple assays will be developed for cost-effective detection of target proteoforms for early detection of cancer.

Overall conduct of the study is the responsibility of the recruiting facilities/physicians. LifeStory Health provides operational oversight. The Baylor Scott and White Research Division (BSW) is responsible for oversight of the Regional Centers. LifeStory Health is responsible for data collection,management and analysis. Study patient safety and study performance are monitored by BSW. This study is being conducted with LifeStory Health and principal investigator, Anna Villarreal, CEO and Founder of LifeStory Health Inc.This randomized, double blind, controlled trial will enroll 60 patients.

ELIGIBILITY:
Inclusion Criteria:

* are 18 years or older

  * are either healthy or have a recent diagnosis of breast, endometrial or lung cancer and have not yet begun treatment (your doctor will provide the stage of cancer at time of enrollment)
  * are willing and able to comply with the study requirements
  * have a negative pregnancy test prior to enrolling in this study
  * Have provided all current medication usage and accurately reported disease history (both current and past) and completed the health profile provided at time of enrollment
* currently menstruating

Exclusion Criteria:

* have a generalized infection (bacterial, viral or fungal), or obvious localized infections in the vaginal area
* have any active sexually transmitted diseases•if you become pregnant while on the study, you must withdraw from the study.
* have received an investigational drug within four weeks prior to the study or who plan to use other investigational drugs duringthis study.
* have severe medical condition(s) that in the view of the investigator prohibits participation in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Three sites will serve as participant recruitment:
  Baylor Scott & White Medical Center - Hillcrest Baylor Scott & White Medical Center - Round Rock Scott & White Medical Center - Temple
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-05-15 (Estimated); Primary Completion 2019-11-01 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Use UPLC UHR-MS and UPLC IM-MS to confirm previous findings of unique signatures in menstrual blood. The sponsor will additionally measure and new biomarkers in menstrual blood for early detection of breast, endometrial, and lung cancers. | 8 weeks
  UHR-MS and IM-MS, in parallel, for proteomics analysis of MB. These two approaches offer complementary advantages for comprehensive proteomic studies and assure detection of low abundance and post-translationally modified proteins in complex mixtures.

CONTACTS AND LOCATIONS:
Locations (1):
- Vasicek Cancer Treatment Center, Temple, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes